CLINICAL TRIAL: NCT00447616
Title: Prostatectomy Database
Brief Title: Prostatectomy Prospective Database
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Kenneth Peters, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2003-214
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of establishing the database is to evaluate the effects of surgical removal of the prostate (prostatectomy) and cryosurgery on prostate cancer, quality of life, and overall health.

DETAILED DESCRIPTION:
The purpose of establishing the database is to evaluate the effects of surgical removal of the prostate (prostatectomy) and cryosurgery on prostate cancer, quality of life, and overall health. Participation in the study will allow collection of medical information related to prostate cancer treatment from hospital and doctor's office records. Questionnaires will be completed reflecting bladder, bowel, and sexual function, and quality of life at three, six, twelve, eighteen, and twenty-four months after surgery, and yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* males greater than 18 years of age
* patients having prostatectomy or cryosurgery for the treatment of prostate cancer at William Beaumont Hospital.

Exclusion Criteria:

* dementia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having prostatectomy or cryosurgery for the treatment of prostate cancer at William Beaumont Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 896 (Actual)
Dates: Start 2003-10; Primary Completion 2015-04-07 (Actual); Study Completion 2015-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No